CLINICAL TRIAL: NCT00389272
Title: Adding a Second Drug for Febrile Children Treated With Acetaminophen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 53/05
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2006-10

CONDITIONS: Fever
MeSH Terms: conditions — Fever | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Ibuprofen, acetaminophen

SUMMARY:
Fever is one of the most common symptoms in pediatrics and one of the most common reasons for visits in pediatricians' office and pediatric emergency departments. Many parents consider fever to be the most terrifying symptom.

Acetaminophen and ibuprofen are both effective and safe treatments for febrile children. In order to achieve better temperature control and to avoid toxicity it has been suggested to treat febrile children with alternating doses of acetaminophen and ibuprofen. Surveys in the USA and Spain found that this practice is very common. However, The safety and efficacy of such practice was never described.

Hypothesis:

Children who are still febrile after being treated with acetaminophen or ibuprofen will have greater temperature decrement if treated with another drug (acetaminophen for those treated with ibuprofen and ibuprofen for those treated with acetaminophen) than if treated with placebo.

DETAILED DESCRIPTION:
Methods:

Design: randomized double blind placebo controlled study. Setting: The ED and pediatric ward of a large University affiliated Hospital

Participants:

Inclusion criteria:

* Age: 6 mo- 4 years
* Rectal temperature > 38.5
* Received 10-15 mg/kg of acetaminophen or 5-10 mg/kg of ibuprofen 1.5 - 3.5 hours before admission to the ED.

Exclusion criteria:

* Received more than 75 mg acetaminophen in the last 24 hours
* Unable to take oral medications
* Hypersensitivity to acetaminophen or ibuprofen
* Varicella
* Renal failure
* Liver disease
* Rectal temperature can't be measured (due to anatomical or medical problem)
* Received both Ibuprofen and acetaminophen in the last 6 hours
* Informed consent could not be granted

Intervention:

Patients will be recruited in the ED and pediatric ward at Assaf Harofeh Medical Center. Legal guardians of eligible patients will be approached for consent. After obtaining informed consent a detailed history regarding the way fever was managed during the current illness will be collected (appendix 1). Patients will be randomized in a ratio of 2:1 (by a computer generated list of random numbers) into one of two groups. Group A will be treated with oral suspension of ibuprofen 10mg/kg (if the patient received acetaminophen at home) or oral suspension of acetaminophen 15 mg/kg (if treated previously with ibuprofen). The second group will be treated with the same amount of oral placebo suspension. The parents and the physician will be blinded to the treatment given. Body departure will be recoded at base line and at 15, 30, 60, 90, 120, 180 minutes after the drug administration. Blood sample for serum concentrations of acetaminophen or/and ibuprofen will be taken at the time of routine blood sampling according to the attending physician decision. Serum concentrations will not be measured if the attending physician decides that blood tests are not indicated.

Primary outcome:

· Maximal change in temperature during the 3-hour period after enrollment.

Secondary endpoints:

* Proportion of patients with a drop of at least 1°C and 2°C in mean temperature at the end of the study (3 hours).
* Decrement in fever at each time point, and the area under the temperature (versus time) curve for each group, calculated using the trapezoidal method. Continuous outcomes
* Proportion of patients with temperature < 38 at the end of the study (3 hours).

ELIGIBILITY:
Inclusion Criteria:

* Age: 6 mo- 4 years
* Rectal temperature > 38.5
* Received 10-15 mg/kg of acetaminophen or 5-10 mg/kg of ibuprofen 1.5 - 3.5 hours before admission to the

Exclusion Criteria:

* Received more than 75 mg acetaminophen in the last 24 hours
* Unable to take oral medications
* Hypersensitivity to acetaminophen or ibuprofen
* Varicella
* Renal failure
* Liver disease
* Rectal temperature can't be measured (due to anatomical or medical problem)
* Received both Ibuprofen and acetaminophen in the last 6 hours
* Informed consent could not be granted

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2005-09; Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Eran Kozer, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Pediatric Emergency Medicine Service, Assaf Harofeh Medical Center, Ẕerifin, Israel